CLINICAL TRIAL: NCT07063901
Title: Multimodal Deep Learning for Predicting Treatment Response to Neoadjuvant Chemoimmunotherapy in Esophageal Cancer
Status: Recruiting | Type: Observational
Sponsor: Central South University (Other)
Responsible Party: Principal Investigator, Chen Chen, Associate Professor, Central South University
Other Study IDs: LYF20250118
Record Dates: First submitted 2025-07-03; First posted 2025-07-14 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-07

CONDITIONS: Esophagus Cancer
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- group 1: pCR: group 1: Pathologic Complete Response
- group 2: Non-pCR: group 2: Non-Pathological Complete Response
- group 3: Non-Favorable Responses: group 3: SD/PD
- group 4: Favorable Response: group 4: Non-SD/PD

SUMMARY:
This observational study aims to investigate a clinical cohort of patients with locally advanced esophageal cancer undergoing neoadjuvant chemoimmunotherapy. By integrating multimodal clinical data-including demographic characteristics, medical history, imaging studies, pathological findings, and laboratory tests-and employing deep learning algorithms, the study seeks to develop predictive models for the early and accurate assessment of treatment response prior to surgery. Specifically, this study focuses on addressing the following key scientific questions:

1. Can multimodal clinical data be used to construct an accurate model for predicting pathological complete response (pCR) following neoadjuvant therapy?
2. Can deep learning models enable early identification of patients with suboptimal response to neoadjuvant therapy, defined as stable disease (SD) or progressive disease (PD), before surgery?

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically confirmed esophageal cancer based on biopsy results;
2. Patients recommended for neoadjuvant chemoimmunotherapy following multidisciplinary team (MDT) discussion or evaluation by thoracic surgery specialists;
3. Patients who received neoadjuvant chemoimmunotherapy;
4. Patients with complete imaging data before and after neoadjuvant treatment.

Exclusion Criteria:

1. Patients deemed eligible for surgery by the thoracic surgery team but who refused surgical treatment;
2. Patients with missing or poor-quality CT images;
3. Patients with concurrent malignancies other than esophageal cancer;
4. Patients with incomplete clinical data.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with esophageal cancer who received neoadjuvant therapy at the Second Xiangya Hospital of Central South University
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
pCR | From enrollment to the end of surgery
  Pathologic Complete Response

SECONDARY OUTCOMES:
Non-Favorable Responses | From enrollment to the end of surgery
  stable disease/progressive disease

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Xiangya Hospital of Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No